CLINICAL TRIAL: NCT01688700
Title: A Prospective, Single Arm, Multicenter, Phase II Study of Nimotuzumab in Combination With Neoadjuvant Chemotherapy for Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Study of Nimotuzumab in Combination With Neoadjuvant Chemotherapy for Resectable Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NimoESCC
Record Dates: First submitted 2012-09-16; First posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Esophageal Squamous Cell Carcinoma Resectable
Keywords: Esophageal Squamous Cell Carcinoma; neoadjuvant therapy; Nimotuzumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nimotuzumab plus chemotherapy (Experimental)
  Interventions: Drug: Nimotuzumab combined with paclitaxel and cisplatin

INTERVENTIONS:
Drug: Nimotuzumab combined with paclitaxel and cisplatin — Nimotuzumab: 200mg, IV once a week for 6 weeks during chemotherapy (days 1,8,15,22,29,36).
  Cisplatin: 75mg/m2,IV on days 1，22
  paclitaxel: 90mg/m2, IV on days 1,8,22,29.
  patients will receive radical operation 4-6 weeks after Neoadjuvant therapy.

SUMMARY:
A higher percentage of radical resection is reported in studies using neoadjuvant chemotherapy followed by surgery versus surgery alone for esophageal cancer. And neoadjuvant chemotherapy may improve overall survival after surgical resection. Nimotuzumab is a humanized monoclonal antibody against epidermal growth factor receptor (EGFR). The concurrent trial is a clinical phase II trial designed to assess the efficacy of the combination of Nimotuzumab administered concurrently with neoadjuvant chemotherapy in patients with resectable Esophageal Squamous Cell Carcinoma, and to further investigate its side-effect and toxicity

DETAILED DESCRIPTION:
A surgical resection is currently the preferred treatment for esophageal cancer if the tumor is considered to be resectable without evidence of distant metastases. A higher percentage of radical resection is reported in studies using neoadjuvant chemotherapy followed by surgery versus surgery alone. The neoadjuvant chemotherapy may improve overall survival. Neoadjuvant chemotherapy with administrations of paclitaxel combined with cisplatin or carboplatin has shown effectively. Nimotuzumab is a humanized monoclonal antibody against epidermal growth factor receptor (EGFR). The clinical phase I study of the combination of Nimotuzumab administered concurrently with chemo-irradiation in patients with local advanced esophageal squamous cell carcinoma has shown the safety and the potential efficacy of Nimotuzumab. The concurrent trial is a clinical phase II trial designed to assess the efficacy of the combination of Nimotuzumab administered concurrently with neoadjuvant chemotherapy in patients with resectable Esophageal Squamous Cell Carcinoma, and to further investigate its side-effect and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologic diagnosis of Esophageal squamous cell carcinoma
* ECOG performance status 0-2
* Age:18-70 years
* Joined the study voluntarily and signed informed consent form
* Patients must not have received any prior anticancer therapy
* Resectable disease, Stage IIA-IIIC, T2N0M0-T3N1M0（AJCC 2009）
* Target lesions can be measured according to RECIST criteria
* No serious system dysfunction and immuno-deficiency, Adequate organ function including the following: Hemoglobin ≥9 g/dL, WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L, platelet count ≥100x 109/L, TBIL<1.5 x ULN, ALT and AST ≦ 2.5 x ULN, creatinine ≦ 1.5 x ULN
* Use of an effective contraceptive for adults to prevent pregnancy
* Life expectancy of more than 3 months

Exclusion Criteria:

* Not suitable to surgery
* cervical Esophageal Carcinoma(distance of incisor tooth<19cm)
* early Esophageal Carcinoma(Stage I)
* complete esophageal obstruction，Esophageal perforation or hematemesis
* other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ
* pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior 11、 History of serious allergic or castor oil allergy 12、 Patients who are not suitable to participate in the trial according to researchers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Pathology complete remission rate | 1 year
  Pathology complete remission rate is the primary outcome measure.

SECONDARY OUTCOMES:
R0 resection rate | 1 year
objective response rate | 1 year
  Objective response rate of neoadjuvant chemotherapy will be assessed.
overall survival | 5 years
tolerability and safety | 2 years
  number of adverse events such as leucopenia ,rash,diarrhea and so on
Quality of life | 5 years
  Quality of life of patients will be evaluated during and after therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China